CLINICAL TRIAL: NCT06609421
Title: Observational Cohort Study of Oocyte Physiology in Discarded Samples of Patients Undergoing IVF
Brief Title: Egg Quality Assessment
Status: Suspended | Type: Observational
Why Stopped: End of collaboration with research site.
Sponsor: Ovom Care GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: 340652
Record Dates: First submitted 2024-09-22; First posted 2024-09-24 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Infertility (IVF Patients); Ovarian Aging; IVF
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Discarded, unfertilised oocytes and follicular fluid collected during routine oocyte retrieval
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Control Group: Women undergoing in-vitro fertilisation (IVF) with male factor diagnoses.
  Interventions: Other: Informative Appointment
- Case Group: Women undergoing IVF with a diagnosis other than male factor.
  Interventions: Other: Informative Appointment

INTERVENTIONS:
Other: Informative Appointment — The only intervention involving the participants is non-clinical, which is an extra 30-minute informative telephone appointment added to the standard care consultation schedule of interested IVF patients where they will be presented with a digital consent PDF form to sign by a study nurse or clinically trained research personnel. Participants will be in the study for 24-30 months. During this time their discarded, unfertilised oocytes and follicular fluid collected during routine oocyte retrieval along with information from their electronic medical records will be collected and analysed.

SUMMARY:
The goal of this observational study is to learn about egg physiology in humans.

The main question it aims to answer is if there is an association between egg physiology and egg quality.

Discarded, unfertilised eggs and follicular fluid collected during routine egg retrieval from participants undergoing in vitro fertilisation (IVF) as part of their regular medical care along with information from participants' electronic medical records will be collected and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing in vitro fertilisation treatment or egg freezing

Exclusion Criteria:

* No discarded, unfertilised eggs for collection

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with uteri experiencing infertility issues requiring assisted reproduction via in vitro fertilisation (IVF)/intracytoplasmic sperm injection (ICSI) or undergoing elective egg freezing.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial physiology in the oocytes | Baseline time of observation which lasts between 1 and 5 hours

SECONDARY OUTCOMES:
Comparison of oocyte mitochondrial physiology results to clinical outcomes to assess correlation (or lack thereof) | As the data becomes available over the course of the participants' medical treatment. E.g. From enrolment until birth of an infant

CONTACTS AND LOCATIONS:
Locations (1):
- Avenues Clinic, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brayboy LM, Oulhen N, Witmyer J, Robins J, Carson S, Wessel GM. Multidrug-resistant transport activity protects oocytes from chemotherapeutic agents and changes during oocyte maturation. Fertil Steril. 2013 Nov;100(5):1428-35. doi: 10.1016/j.fertnstert.2013.07.002. Epub 2013 Aug 13. PMID 23953328